CLINICAL TRIAL: NCT04459793
Title: The Danish Occupational Medicine Cohort - Long-term Prognosis for Patients With Work-related Disorders
Acronym: PRORISK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Regional Hospital West Jutland (Other)
Collaborators: Aarhus University Hospital Skejby (Other); University of Aarhus (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, David H Christiansen, Associate Professor, Regional Hospital West Jutland
Other Study IDs: DST7055
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Work-Related Condition
Keywords: Prognosis; Work-related disorders; Occupational medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Each year about 10.000 patients are referred due to suspected work-related disorders to the Danish departments of occupational medicine. In Denmark and internationally there is a lack of follow-up studies investigating the long-term prognosis of employees with work-related disorders. To facilitate long-term prognostic studies for work-related conditions a Danish Occupational Medicine Cohort has been established through the Danish population registers.

DETAILED DESCRIPTION:
Danish departments of occupational medicine examine around 10,000 patients each year referred due to suspected work-related disorders. In Denmark and internationally there is a lack of follow-up studies investigating the long-term prognosis of employees with work-related disorders. The purpose of this cohort is to facilitate long-term prognostic studies for conditions such as mental or musculoskeletal disorders.

The Danish Occupational Medicine cohort has been created through The Danish National Patient Register and comprises all patients seen in Danish Departments of Occupational Medicine from 2000-2018 (N=145.521). Numerous register data are included in the database from five years prior to time of inclusion until 2018. Examples of register data are; information on work, sickness absence and disability as well as number and type of contacts to health services, use of medication, income, education, type of occupation, social status, death and cause of death. Job Exposure Matrices (JEMs) on physical and psychosocial work exposure, life styles and other matrices are also available. The cohort will be updated with new patients and register data regularly.

ELIGIBILITY:
Inclusion Criteria:

* A record of contact at Danish departments of occupational medicine with a relevant primary or secondary diagnosis according to the International Classification of Diseases, 10th revision.

Exclusion Criteria:

* No record of contact or only a record of referral without subsequent records of relevant primary or secondary diagnosis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort was created through The Danish National Patient Register and comprises all patients seen in Danish Departments of Occupational Medicine from 2000-2018 (N= 145.521). Numerous register data are included in the database from five years prior to time of inclusion until 2018. The cohort will be updated with new patients and register data regularly.
Sampling Method: Non-Probability Sample
Enrollment: 145521 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Annual work participation score | 5 years
  Work participation score is defined as number of weeks of employment relative to the total sum of number of weeks of employment plus number of weeks on temporary or permanent health related public compensation as registered by the Danish National Register on Public Transfer Payments register (DREAM).
Annual health care utilization | 5 years
  Primary and secondary Health care contacts - includes all face to face contacts from the Danish National Health Service Register and Danish National Patient Register

CONTACTS AND LOCATIONS:
Overall Officials: David H Christiansen, Principal Investigator — Occupational Medicine, Regional Hospital Herning
Locations (1):
- David H Christiansen, Herning, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Persson ML, Willert MV, Kyndi M, Dalgaard VL. Work participation and disability pension after work-related PTSD: trajectories and impact of occupation. Occup Environ Med. 2026 Feb 3:oemed-2025-110412. doi: 10.1136/oemed-2025-110412. Online ahead of print. PMID 41633844
- [Derived] Willert MV, Christiansen DH, Dalgaard L, Vestergaard JM, Andersen JH, Kyndi M. Developing prognostic models for health care utilization in patients with work-related mental health problems. BMC Health Serv Res. 2023 Aug 7;23(1):834. doi: 10.1186/s12913-023-09802-z. PMID 37550656